CLINICAL TRIAL: NCT05214651
Title: A Clinical Research on Arthroscopic Repair of Massive-large Rotator Cuff Tears With a Novel Inner Fixation Technique
Brief Title: A Clinical Research on Repair of Massive-large Rotator Cuff Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2021389
Record Dates: First submitted 2021-12-29; First posted 2022-01-31 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tears
Keywords: novel double row technique; suture bridge double row technique; massive-large rotator cuff tears; retear rate
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- novel double row group (Experimental): This is the experimental group, and 26 participants will be enrolled, a novel double row technique will be using to repair the large - massive rotator cuff tears in in this group.
  Interventions: Procedure: novel double row
- suture bridge double row group (Active Comparator): This is the control group, and 26 participants will be enrolled, a suture bridge double row technique will be using to repair the large - massive rotator cuff tears in in this group in routine.
  Interventions: Procedure: suture bridge double row

INTERVENTIONS:
Procedure: novel double row — The large - massive rotator cuff tears in in this group will be treated using a novel double row repairing techniques.
  Arms: novel double row group
Procedure: suture bridge double row — The large - massive rotator cuff tears in in this group will be treated using a suture bridge double row repairing techniques.
  Arms: suture bridge double row group

SUMMARY:
The study is designed as a randomized controlled trial, a total of 52 participants with large - massive rotator cuff tears will be prospectively enrolled and randomly divided into 2 groups according to the applied repairing technique: novel double row technique group and suture bridge double row technique group. The functional outcome was measured at the preoperatively, 3, 6, 12 and 24 months postoperatively, using the visual analog scale (VAS) for pain, active and passive ROM, Constant score, American Shoulder and Elbow Surgeons (ASES) score, and University of California Los Angeles shoulder score (UCLA). The anatomic outcome was evaluated using magnetic resonance imaging at 3, 6, 12 and 24 months postoperatively. The clinical results were compared between the novel double row technique group and suture bridge double row technique group.

DETAILED DESCRIPTION:
The purpose of this study is to compare a novel double row technique with suture bridge double row technique in the arthroscopic repair of massive-large rotator cuff tears clinically. The study is designed as a randomized controlled trial. A total of 52 participants with large - massive rotator cuff tears will be prospectively enrolled and randomly divided into 2 groups according to the applied repairing technique: novel double row technique group and suture bridge double row technique group.

The investigators prospectively enrolled participants who met the following inclusion criteria: preoperative magnetic resonance imaging (MRI) diagnosis of a large - massive sized rotator cuff tear (>3cm), which was confirmed during operation; chronic tear; older than 17 years and younger than 75 years; without surgical contraindications and willing to participate. The investigators excluded patients with poor quality rotator cuff and irreparable tear; severe glenohumeral arthritis; previous shoulder surgery; accompanied by dislocation or fracture of shoulder; refusal to participate.

Each participant, assigned using a randomization table, was assessed by a clinical researcher, who was blinded to the grouping, at the following time points: preoperatively; 3, 6, 12 and 24 months postoperatively. The visual analog scale (VAS) for pain, active and passive ROM, and functional scores were assessed at each time point. The functional scores including the Constant score, American Shoulder and Elbow Surgeons (ASES) score, and University of California Los Angeles shoulder score (UCLA). Anatomic healing was evaluated using MRI at 3, 6, 12 and 24 months postoperatively. An experienced musculoskeletal radiologist interpreted the MRI and determined the healing failure rate. On the basis of the MRI findings, type IV or V of the Sugaya classification was regarded as healing failure.

Based on the previous study, the retear rate of large to massive rotator cuff tears treated with suture bridge double row technique was assumed to be 28.3%. Based on the investigators' previous clinical data on large to massive rotator cuff tears, it is assumed that the retear rate of large to massive rotator cuff tears treated with novel double row technique is 1.0%.

Differences in primary end points between the two groups were analyzed using chi-square tests. Set α=0.05, power is 0.80, the sample ratio of the two groups was 1:1. The sample size was estimated with PASS 15.0. A total of 46 patients, with 23 in each group, had sufficient power to detect statistical differences between groups. In consideration of the uncertainty of the effect and the possible loss of follow-up, the design effect was assumed to 10%. Therefore, the total sample size of this study should be more than 46÷90%≈51. To facilitate randomization, the sample size was determined to be 52 patients, with 26 patients in each group.

Variables such as age, sex, tear size, and functional scores were analyzed, and their mean values were obtained. Continuous data were presented as the mean ± SD, and were analyzed using the independent t test. The retear rates between the two groups were analyzed using chi-square tests. Differences in values between the 2 groups were set at P < .05 to be statistically significant. All statistical analyses were performed using SPSS version 15.0

ELIGIBILITY:
Inclusion Criteria:

* preoperative magnetic resonance imaging (MRI) diagnosis of a large - massive sized rotator cuff tear (>3cm), which was confirmed during operation
* chronic tear
* older than 17 years and younger than 75 years
* without surgical contraindications and willing to participate

Exclusion Criteria:

* poor quality rotator cuff and irreparable tear
* severe glenohumeral arthritis
* previous shoulder surgery
* accompanied by dislocation or fracture of shoulder
* refusal to participate

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The retear rate of large to massive rotator cuff tears | The incidence of retear during 24 months postoperatively
  This study statistically compared the retear rate of large to massive rotator cuff tears treated with suture bridge double row technique with that treated with novel double row technique.

SECONDARY OUTCOMES:
functional scores of the shoulder | functional scores of the shoulder were assessed at following time points: preoperatively; 3, 6, 12 and 24 months postoperatively
  This study statistically compared the functional scores of the shoulder of large to massive rotator cuff tears treated with suture bridge double row technique with that treated with novel double row technique. The functional scores including the Constant score (0-100), American Shoulder and Elbow Surgeons score (0-100), and University of California Los Angeles shoulder score (2-35). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, M.D., Principal Investigator — Institute of Sports Medicine, Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No